CLINICAL TRIAL: NCT00130026
Title: A Prospective, Randomized, Double-blind, Placebo-controlled Study of Caffeine in the Prevention of Post-operative Nausea and Vomiting in Patients Undergoing Ambulatory Surgery Under General Anesthesia
Brief Title: Caffeine in the Prevention of Post-operative Nausea and Vomiting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Richard A. Steinbrook, Associate Professor of Anaesthesia, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2004P000210
Record Dates: First submitted 2005-08-11; First posted 2005-08-15 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Postoperative Nausea and Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Caffeine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- I (Placebo Comparator): Saline placebo
  Interventions: Drug: Caffeine

INTERVENTIONS:
Drug: Caffeine — 500 mg IV

SUMMARY:
The objective of this study is to determine if caffeine 500 mg intravenously is efficacious when added to standard anti-emetic prophylaxis in the prevention of post-operative nausea and vomiting (PONV) in patients undergoing ambulatory surgery under general anesthesia.

DETAILED DESCRIPTION:
This is a prospective, randomized, double-blind, placebo-controlled study of caffeine, 500 mg, intravenously, in addition to standard anti-emetic prophylaxis, in the prevention of post-operative nausea and vomiting in patients undergoing ambulatory surgery under general anesthesia.

Consenting patients will be randomized to receive either a single dose of caffeine, 500 mg, or saline placebo, administered as a single IV dose approximately 15 minutes before emergence from anesthesia. All patients will receive our customary anti-emetic prophylaxis, determined by four major risk factors for PONV: female gender, nonsmoking status, history of PONV or motion sickness, and perioperative opioid use. Patients at low risk for PONV (no risk factors) will receive no prophylaxis; patients at moderate risk for PONV (1 or 2 risk factors) will receive dexamethasone 8 mg at induction plus dolasetron 12.5 mg approximately 15 min before the end of anesthesia; patients at high risk for PONV (3 or 4 risk factors) will receive the same treatment as those at moderate risk, plus additional prophylaxis at the discretion of the attending anesthesiologist (e.g., scopolamine patch, metoclopramide 10 mg IV, or other standard drugs).

Postoperatively, the presence of PONV will be recorded. If rescue medication is used, the amount and time of administration will be recorded. The length of stay in the PACU (Phase I and Phase II) will be recorded. Patients will be asked to report any headache, and to rate their nausea, pain, alertness, fatigue, and overall satisfaction in the PACU, and again by phone 24 hours postoperatively. Amount of pain medication utilized in the PACU will also be measured.

ELIGIBILITY:
Inclusion Criteria:

* Patient having ambulatory surgery
* Patient receiving general anesthesia

Exclusion Criteria:

* Patient is not willing to sign informed consent
* Patient does not speak or understand sufficient English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2005-03; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Complete response (no PONV and no use of rescue medication) during the first 24 hours following anesthesia | 1-24 hours post-operatively

SECONDARY OUTCOMES:
Nausea during the first 24 hours following anesthesia | 1-24 hours post-operatively
Vomiting during the first 24 hours following anesthesia | 1-24 hours post-operatively
Proportion of patients who use rescue medication during the first 24 hours following anesthesia | 1-24 hours post-operatively
Post Anesthesia Care Unit (PACU) length of stay (Phase I, Phase II) | hours post-operatively
Incidence of headache | 1-24 hours post-operatively
Degree of fatigue | 1-24 hours post-operatively
Overall satisfaction | 1-24 hours post-operatively
Alertness | 1-24 hours post-operatively
Admissions | 1-24 hours post-operatively
Amount of pain medication required | 1-24 hours post-operatively

CONTACTS AND LOCATIONS:
Overall Officials: Richard A Steinbrook, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States